CLINICAL TRIAL: NCT03365206
Title: Oral Health Knowledge and Practice Among 15-17 Year Old Adolescents.
Brief Title: Oral Health Among Adolescents.
Acronym: Oral health
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0414
Record Dates: First submitted 2017-12-01; First posted 2017-12-07 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Dental Consultation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire on practices and knowledge in terms of oral hygiene — Questionnaire on practices and knowledge in terms of oral hygiene during a dental consultation

SUMMARY:
The aim of this study is to identify the knowledge and behavior on dental health and hygiene among adolescents. In most cases, the investigators know tooth decay can be prevented and reversed at an early stage by observing good oral hygiene. Few studies have been done among adolescents.

This study could justify the implementation of public health actions in terms of prevention.

ELIGIBILITY:
Inclusion criteria:

* All adolescents who speek french
* Good general health
* Educated

Exclusion criteria:

* Patients with significant pathologies
* Patients unable to answer questions.
* Non-cooperative patient

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 15 - 17 year old adolescents
Sampling Method: Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
knowledge of oral prevention | 1 day
  Questionnaire on knowledge of oral prevention

OTHER OUTCOMES:
oral habits | 1 day
  Questionnaire on oral habits

CONTACTS AND LOCATIONS:
Overall Officials: Camille INQUIMBERT, PhD student, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC